CLINICAL TRIAL: NCT03767348
Title: An Open-Label, Multicenter, Phase 1/2 Study of RP1 as a Single Agent and in Combination With PD1 Blockade in Patients With Solid Tumors [IGNYTE]
Brief Title: Study of RP1 Monotherapy and RP1 in Combination With Nivolumab (IGNYTE)
Acronym: IGNYTE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Replimune Inc. (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RPL-001-16; 2016-004548-12 (EudraCT Number); 2024-511728-15-00 (EU CTIS Number)
Record Dates: First submitted 2018-12-05; First posted 2018-12-06 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC); Microsatellite Instability-High (MSI-H); Non-melanoma Skin Cancer (NMSC); Cutaneous Melanoma
Keywords: RPL-001-16; Stage IIIb-IV Unresectable Melanoma; Non-melanoma Skin Cancer; Mismatch Repair Deficient (dMMR) Solid Tumors
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Melanoma; Turcot syndrome | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Dose escalation of RP1 by intratumoral (IT) injection in superficial tumors (Experimental): anti-PD-1 monoclonal antibody
  Interventions: Biological: RP1
- Dose escalation of RP1 by intratumoral (IT) injection in deep/visceral tumors (Experimental): Dose escalation of RP1 alone in 3 cohorts with IT injections in superficial tumors
  Interventions: Biological: RP1
- Dose expansion of RP1 and nivolumab (IV) in superficial tumors (Experimental): Dose escalation of RP1 alone in 3 cohorts with IT injections in superficial tumors
  Interventions: Biological: RP1; Biological: nivolumab
- Dose expansion of RP1 and nivolumab (IV) in deep/visceral tumors (Experimental): Doses of RP1 (IT) in deep/visceral tumors with nivolumab (IV)
  Interventions: Biological: RP1; Biological: nivolumab
- RP1 (IT) and nivolumab (IV) in melanoma (Experimental): Doses of RP1 (IT) in superficial or deep tumors with nivolumab (IV) in subjects with melanoma
  Interventions: Biological: RP1; Biological: nivolumab
- RP1 (IT) and nivolumab (IV) in MSI-H/dMMR solid tumors (Experimental): Doses of RP1 (IT) in superficial or deep tumors with nivolumab (IV) in subjects with MSI-H or dMMR solid tumors
  Interventions: Biological: RP1; Biological: nivolumab
- RP1 (IT) and nivolumab (IV) in NMSC (Experimental): Doses of RP1 (IT) in superficial or deep tumors with nivolumab (IV) in subjects with non-melanoma skin cancer
  Interventions: Biological: RP1; Biological: nivolumab
- RP1(IT) and nivolumab (IV) in anti-PD1 Failed Cutaneous Melanoma (Experimental): Doses of RP1 (IT) in superficial or deep tumors with nivolumab (IV) in subjects with cutaneous melanoma who have been previously treated with anti-PD1 therapy
  Interventions: Biological: RP1; Biological: nivolumab
- RP1(IT) and nivolumab (IV) in anti-PD1/PD-L1 Failed NMSC (Experimental): Doses of RP1 (IT) in superficial or deep tumors with nivolumab (IV) in subjects with non-melanoma skin cancer who have been previously treated with anti-PD1/PD-L1 therapy
  Interventions: Biological: RP1; Biological: nivolumab
- RP1(IT) and nivolumab (IV) in anti-PD1/PD-L1 Failed NSCLC (Experimental): Doses of RP1 (IT) in superficial or deep tumors with nivolumab (IV) in subjects with non small cell lung cancer who have been previously treated with anti-PD1/PD-L1 therapy
  Interventions: Biological: RP1; Biological: nivolumab

INTERVENTIONS:
Biological: RP1 — Genetically modified herpes simplex type 1 virus
Biological: nivolumab — anti-PD-1 monoclonal antibody
  Other Names: Opdivo
  Arms: Dose expansion of RP1 and nivolumab (IV) in deep/visceral tumors; Dose expansion of RP1 and nivolumab (IV) in superficial tumors; RP1 (IT) and nivolumab (IV) in MSI-H/dMMR solid tumors; RP1 (IT) and nivolumab (IV) in NMSC; RP1 (IT) and nivolumab (IV) in melanoma; RP1(IT) and nivolumab (IV) in anti-PD1 Failed Cutaneous Melanoma; RP1(IT) and nivolumab (IV) in anti-PD1/PD-L1 Failed NMSC; RP1(IT) and nivolumab (IV) in anti-PD1/PD-L1 Failed NSCLC

SUMMARY:
The Phase 2 study is a multicenter, open-label study of RP1 to further investigate safety and to estimate the efficacy of RP1 at the RP2D in combination with nivolumab in patients with Stage IIIb-IV unresectable melanoma, microsatellite instability-high (MSI-H) or mismatch repair deficient (dMMR) solid tumors, non-melanoma skin cancer (NMSC), and non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Key Inclusion Criteria:

* Have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1.
* At least one measurable and injectable lesion
* Have provided a former tumor pathology specimen or be willing to supply a new tumor sample from a biopsy
* Have a predicted life expectancy of ≥ 3 months
* Measurable disease, according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria
* Subjects with MSI-H or dMMR tumors: has diagnosis of MSI-H or metatstatic dMMR tumor (according to protocol definition) who has progressed on prior anti-PD1/PD-L1 therapy.
* Subjects with NMSC: has diagnosis of locally advanced or metastatic NMSC that are not considered treatable by surgery including basal cell carcinoma, cutaneous squamous cell carcinoma, basosquamous carcinoma, Merkel cell carcinoma and other non-melanoma skin cancers (per protocol). Patients must have received 8 weeks of anti-PD1/PD-L1 as their last line of therapy and progressed while on treatment.
* Subjects with anti-PD1 failed cutaneous melanoma: has confirmed progressive disease while on anti-PD1 treatment for at least 8 weeks and documented BRAF mutation status
* Subjects with anti-PD1 failed NSCLC: must have failed prior treatment, including PD1/PD-L1 directed therapy administered either as monotherapy or in combination with platinum-based chemotherapy or anti-CTLA-4. The most recent treatment given must have included an anti-PD1/PD-L1 directed therapy with radiologic disease progression on or after treatment.

Key Exclusion Criteria:

* Prior treatment with an oncolytic therapy
* History of viral infections according to the protocol
* Prior complications with herpes infections
* Chronic use of anti-virals
* Uncontrolled/untreated brain metastasis
* History of interstitial lung disease
* History of non-infectious pneumonitis
* History of clinically significant cardiovascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2017-09-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of adverse events (AEs) | 26 months
  Percentage of subjects with adverse events (AEs)
Percentage of serious adverse events (SAEs) | 26 months
  Percentage of subjects with serious adverse events (SAEs)
Percentage of dose limiting toxicities (DLTs) | 26 months
  Percentage of subjects with dose limiting toxicities (DLTs)
Percentage of overall response rate (ORR) | 26 months
  Percentage of overall response rate (ORR) for all participants
Maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) of RP1 | 20 weeks
  Assess the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) of RP1 based on the safety and response data collected during Phase 1 Escalation

SECONDARY OUTCOMES:
Percentage of biologic activity | 20 weeks
  Percentage of subjects with biological activity determined by tumor biopsies and biomarker data
Percentage subjects with detectable RP1 | 20 weeks
  Data gathered from blood, urine, swabs of injection site, dressings, and oral mucosa to determine the shedding and biodistribution of RP1
Percentage of complete response (CR) | 26 months
  Percentage of subjects with a complete response (CR)
Median duration of response | 26 months
  Median duration of response of subjects
Median progression-free survival | 26 months
  Median duration of progression-free survival of subjects
Median overall survival | 26 months
  Median overall survival rate of subjects

CONTACTS AND LOCATIONS:
Overall Officials: Jeannie Hou, MD, Study Director — Replimune Inc.
Locations (51):
- United States (26):
  - University of Birmingham Alabama, Birmingham, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic, Phoenix, Arizona
  - Carti Cancer Center, Little Rock, Arkansas
  - UC San Diego, La Jolla, California
  - University of Southern California, Los Angeles, California
  - UCLA, Los Angeles, California
  - University of California, Irvine, Orange, California
  - University of California- San Francisco, San Francisco, California
  - Sylvester Comprehensive Cancer Center- University of Miami, Miami, Florida
  - University of Iowa-Cancer Center Research, Iowa City, Iowa
  - James Graham Brown Cancer Center- University of Louisville, Louisville, Kentucky
  - Mayo Clinic, Rochester, Minnesota
  - New York University Clinical Cancer Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Duke Cancer Center, Durham, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - MUSC Health, Charleston, South Carolina
  - West Cancer Center, Germantown, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Eccles Outpatient Care Center- Oncology Clinical Trials, Murray, Utah
  - Intermountain Cancer Center- Saint George Cancer Center, St. George, Utah
  - Seattle Cancer Care Alliance- University of Washington, Seattle, Washington
  - University of Wisconsin-Carbone Cancer Center, Madison, Wisconsin
- France (8):
  - CHU Besancon - Hopital Jean Minjoz, Besançon
  - Institut Bergonié, Bordeaux
  - CHU Dijon, Dijon
  - Centre Léon Bérard Lyon, Lyon
  - Service de Dermatologie et Cancerologie Cutanee Hopital de la Timone, Marseille
  - CHU de Nice Hôpital l'Archet, Nice
  - Hôpital Saint Louis APHP, Paris
  - Institut Gustave Roussy, Villejuif
- Germany (4):
  - Charité (Campus Benjamin Franklin), Berlin
  - University Hospital Essen, Klinik für Dermatologie, Essen
  - University of Kiel (UKSH), Dep. of Dermatology, Kiel
  - Uniklinik Marburg, Marburg
- Spain (7):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - Clínica Universidad de Navarra (Madrid), Madrid
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Clinica Universitaria de Navarra, Pamplona
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital General Universitario de Valencia, Valencia
- United Kingdom (6):
  - University of Leeds- Teaching Hospital, Leeds, England
  - Oxford University Hospitals NHS Trust, Oxford, Oxfordshire
  - Beatson West of Scotland Cancer Center, Glasgow, Scotland
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Bebington, Wirral
  - Royal Marsden Hospital, London
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong MK, Milhem MM, Sacco JJ, Michels J, In GK, Munoz Couselo E, Schadendorf D, Beasley GM, Niu J, Chmielowski B, Wise-Draper TM, Bowles TL, Tsai KK, Lebbe C, Gaudy-Marqueste C, Middleton MR, Skolariki A, Samson A, Chesney JA, VanderWalde AM, Zakharia Y, Harrington KJ, Appleton E, Bommareddy PK, Zhu J, Viana M, Hou JW, Coffin RS, Robert C. RP1 Combined With Nivolumab in Advanced Anti-PD-1-Failed Melanoma (IGNYTE). J Clin Oncol. 2025 Nov 20;43(33):3589-3599. doi: 10.1200/JCO-25-01346. Epub 2025 Jul 8. PMID 40627813
- [Derived] Thomas S, Kuncheria L, Roulstone V, Kyula JN, Mansfield D, Bommareddy PK, Smith H, Kaufman HL, Harrington KJ, Coffin RS. Development of a new fusion-enhanced oncolytic immunotherapy platform based on herpes simplex virus type 1. J Immunother Cancer. 2019 Aug 10;7(1):214. doi: 10.1186/s40425-019-0682-1. PMID 31399043